CLINICAL TRIAL: NCT01501578
Title: Phenotype of Pulmonary Fibrosis Associated With a Mutation of Telomerase
Brief Title: Pulmonary Fibrosis and Telomerase Mutation Study
Status: Completed | Type: Observational
Sponsor: Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires (Other)
Collaborators: Bichat Hospital (Other)
Responsible Party: Principal Investigator, Vincent COTTIN, Principal Investigator, Groupe d'Etudes et de Recherche sur les Maladies Orphelines Pulmonaires
Other Study IDs: GERMOP-004
Record Dates: First submitted 2011-12-13; First posted 2011-12-29 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Fibrosis
Keywords: Pulmonary fibrosis; Telomerase mutation
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — one blood sample is collected for genetic analysis of telomerase mutation
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- telomerase mutation: Patients with interstitial lung disease and telomerase mutation
- control: Patients with idiopathic pulmonary fibrosis and without telomerase mutation

SUMMARY:
This study is an observational and retrospective study of patients with pulmonary fibrosis associated or not with telomerase mutation.

The purpose of this study is to describe in detail the cases with telomerase mutation in terms of features on CT scan, respiratory function and evolution, in comparison to control subjects with idiopathic pulmonary fibrosis and no telomerase mutation identified or family history.

DETAILED DESCRIPTION:
Two "control" subjects will be enrolled for one subject with telomerase mutation.

The data are all the results of investigations conducted for the diagnosis of idiopathic pulmonary fibrosis and during routine follow up of patients.

The CT scans will reviewed centrally to homogenize the description.

ELIGIBILITY:
Inclusion Criteria:

* Diffuse interstitial lung disease on CT scan
* Telomerase mutation analysis

Exclusion Criteria:

* Presence of connective tissue disease, or pneumoconiosis or drug induced lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with pulmonary fibrosis with and without telomerase mutation
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2011-12; Primary Completion 2012-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Description of imaging pattern | at baseline only
  Description of imaging pattern on representative CT scan at diagnosis.

SECONDARY OUTCOMES:
Pathology of the lung | at baseline only
  description of pathological pattern
Pulmonary function tests | from diagnosis to last follow-up, for an average of one year
  analyze the respiratory function

CONTACTS AND LOCATIONS:
Overall Officials: vincent Cottin, MD, Principal Investigator — Hospices civils de Lyon / University Lyon I
Locations (1):
- Louis Pradel Hospital (Bâtiment A4), Lyon, France

IPD SHARING:
Plan to Share IPD: Yes
Under analysis, publication in preparation

REFERENCES:
- See also: website National French Reference Center for rare lung diseases — http://maladies-pulmonaires-rares.fr/